CLINICAL TRIAL: NCT05531422
Title: Effectiveness and Tolerance of Inhaled Fentanyl Aerosol (25µg/Dose) in Chinese Patients With BTcP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ZK06
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Breakthrough Cancer Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled fentanyl aerosol (Experimental): Participants were randomized to 6 BTP episodes, in which 4 BTP episodes were treated with Inhaled fentanyl aerosol (25 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×25µg) in a random sequence
  Interventions: Drug: Inhaled fentanyl aerosol
- Placebo (Placebo Comparator): Participants were randomized to 6 BTP episodes, in which 2 BTP episodes were treated with placebo (0 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×0µg) in a random sequence
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inhaled fentanyl aerosol — Participants were randomized to 6 BTP episodes, in which 4 BTP episodes were treated with inhaled fentanyl aerosol (with a starting dose of 25 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×25 µg) and 2 BTP episodes with placebo(0 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×0µg) in a random sequence.
  Arms: Inhaled fentanyl aerosol
Drug: Placebo — Participants were randomized to 6 BTP episodes, in which 4 BTP episodes were treated with inhaled fentanyl aerosol (with a starting dose of 25 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×25 µg) and 2 BTP episodes with placebo(0 µg every 4 minutes until adequate pain alleviation. The maximum doses are 6×0µg) in a random sequence.
  Arms: Placebo

SUMMARY:
Breakthrough cancer pain (BTcP) is a common problem in patients with cancer. This is a phase IIa dose-response and safety study of inhaled fentanyl aerosol (25µg/dose) in Chinese patients with breakthrough cancer pain.

DETAILED DESCRIPTION:
Consenting patients who met inclusion and exclusion criteria were allowed to enter the study. The medication for background pain during screening were maintained until the end of the study. Each patient would be treated and observed for 6 episodes of targeted BTcP. Patients were randomly assigned to 1 of the 6 prespecified dose sequences which were established by a computer-generated schedule of active drug and placebo in a 4:2 ratio. All patients and personnel involved with the study (including investigators and investigation site personnel) were blinded to the medication codes.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or above
2. Subjects must be diagnosed with cancer.
3. Subjects must experience persistent pain associated with cancer, and the pain score assessed by NRS should be <4 within 1week before screening.
4. In the past 7 days, the subject must experience an average of 1 to 4 episodes of breakthrough cancer pain per day,The breakthrough cancer pain score should be ≥4 assessed by NRS
5. ECOG status of 0 to 2.
6. Subjects must consent to take adequate contraception during the study and 1 months after the study. Women of childbearing potential must show negative in the pregnancy test before dosing.
7. The subject must be able to understand the requirements of the study and provide a written informed consent.

Exclusion Criteria:

1. History or suspected allergies to fentanyl.
2. HGB < 80 g/L, NEUT ≤1.0 × l09/L, PLT ≤50 × l09/L；ALT and AST higher than 3 times of ULN;total bilirubin and Cr higher than 1.5 times of ULN;PaO2 <95%;FEV1/FVC<70% and FEV1 accounted for less than 80% of the predicted value.
3. Any uncontrolled disease (e.g., severe mental, neurological, infectious, cardiovascular, respiratory and other systemic diseases).
4. Tumor infiltration to central nervous system.
5. Subjects are not able to slef evaluate pain intensity using NRS
6. Receive surgery in past 3 weeks
7. Treatment with any form of radiotherapy winth 1week prior to study entry that could alter pain or response to pain medication.
8. Taking monoamine oxidase inhibitors(MAOIs), CYP3A4 inhibitors or inducers within 14 days of the screening
9. Participated in other clinical trials in past 1months.
10. Pregnancy and breast-feeding women, women of childbearing age ready to conceive, and pregnancy test positive.
11. Other conditions that may affect the informed consent, compliance with the protocol, study results and safety of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
SPID30 | at each episode of breakthrough pain, 30 minutes after first dose of study drug.
  Weighted sum of pain intensity difference at post dose 30 minutes.Pain intensity at each breakthrough pain (BTP) episode at 0 ,4,8,12,16,20 and 30 minutes after first dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain". PID30 is calculated as the difference in pain intensity from time 0 to 30 minutes. A positive value is a decrease (improvement) of the pain.SPID30=PID4*4+PID8*4+PID12*4+PID16*4+PID20*4+PID30*10

SECONDARY OUTCOMES:
Pain intensity at 0, 4,8,12,16,20,30 and 60 minutes post-dose | at each episode of breakthrough pain, 60 minutes after first dose of study drug.
  Pain intensity at each breakthrough pain (BTP) episode at 0 ,4,8,12,16,20, 30 and 60 minutes after first dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain".A positive value is a decrease (improvement) of the pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin R, Song B, Li N, Rong B, Bai J, Liu Y, Wang W, Liu A, Luo S, Liu B, Cheng P, Wu Y, Li Y, Yu X, Liu X, Dai X, Li X, Liu D, Wang J, Huang Y. Efficacy and safety of fentanyl inhalant for the treatment of breakthrough cancer pain: a multicenter, randomized, double-blind, placebo-controlled trial. BMC Palliat Care. 2024 Sep 7;23(1):222. doi: 10.1186/s12904-024-01554-9. PMID 39244530